CLINICAL TRIAL: NCT06041100
Title: Assessing the Long-term Effects of Wearing a Lower-limb Exoskeleton on Physical Activity and Quality of Life in Pre-frail Adults - a Feasibility Study
Brief Title: What Are the Effects of a Bilateral Hip Exoskeleton During Daily Use by 65+ Adults?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Imasen Electrical Industrial Co., Ltd. (Unknown); Aalborg Municipality (Other)
Responsible Party: Principal Investigator, Cristina-Ioana Pirscoveanu, Principal Investigator, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAU2-LBK1083
Record Dates: First submitted 2023-09-01; First posted 2023-09-18 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Pre-frail Senior Adults
Keywords: exoskeleton; aging; walking
MeSH Terms: interventions — Exoskeleton Device

STUDY DESIGN:
Intervention Model Description: All participants will complete three test sessions:
  1. An initial assessment (baseline)
  2. A 4-week assessment and
  3. A 12-week assessment.
  4. Around 8-10 participants will be invited for a follow-up assessment 6-weeks post after the trial has ended.
  All participants will be instructed to wear the device 30 minutes daily during moderate to intensive physical activities. They will be required to provide a weekly overview of their usage and experience with the device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): 30 minutes of daily wearing an exoskeleton for 12-weeks
  Interventions: Device: Exoskeleton

INTERVENTIONS:
Device: Exoskeleton — Use a passive assistive hip exoskeleton (alQ, Imasen Electrical Industrial Co., Ltd.) for 30 minutes daily during moderate to intensive activities over a period of 12-weeks. The exoskeleton is designed to aid hip flexion and as such its primary role is to improve gait by increasing step length and improving speed. The amount of time the exoskeleton has been used will be weekly monitored through phone calls and two gait sessions will be conducted to measure the development.

SUMMARY:
Despite the huge popularity exoskeletons have gained in the past years and the benefits that they have shown to provide to users, there are still many aspects of wearing an exoskeleton that have yet to be determined. Therefore, the main objective of this study is to evaluate the feasibility using the acceptability of incorporating a passive assistive bilateral exoskeleton into the daily routine of pre-frail adults for a duration of 12-weeks. The second aim of the study is to determine whether this effect can be sustained even after a period of 6-weeks following the cessation of usage.

DETAILED DESCRIPTION:
Despite the high benefits of performing physical activity in terms of physical and cognitive function, between 27-38% of Danish older adults do not meet the required physical activity recommendations. Due to the longer life expectancy, the increasingly older population will face gait disorders. These gait disorders will affect their motor and cognitive functions, and impair the performance of daily physical activity and overall quality of life. Frailty is one of the most frequent aging-related deficits observed in older adults, often characterized by three of the following criteria: unintentional weight loss >4.5 kg within the last year, exhaustion, loss or slower mobility, loss of grip strength, and low physical activity. However, pre-frail adults may present some of the aforementioned criteria and a score of ≤5 on the Tilburg Frailty Indicator. Therefore, there is an increasing need to provide the aging population with devices capable of promoting physical activity and independent living. Exoskeletons have been shown to facilitate physical activity in the older adult population by improving metabolic costs, increasing walking speed, and preventing falls. However, whether these benefits are only temporary, or can be maintained over a longer period, remains to be determined. Therefore, it is of pivotal importance to assess the long-term effects of exoskeletons, in terms of mobility, within the older adult population.

The use of external mechanical walking devices started in the late 1890s. However, only in the past two decades have gait-assisting exoskeletons, with increased human performance capability, gained popularity. Exoskeletons have been shown to reduce metabolic cost, and fatigue onset and increase walking velocity. Currently on the market, there are several lower-limb exoskeletons that target older populations and people with gait and neurological disabilities which are designed to enhance walking performance and reduce the muscle activation required during walking activities. Wearing gait-assisting exoskeletons can provide instant ease, delay fatigue onset, increase social engagement, and support rehabilitation to recover normal walking capabilities. The effects of hip exoskeletons have been previously investigated in terms of quality of life and improvement of gait performance. However, the effect of long-term use has yet to be assessed. Hence, this study aims to evaluate the impact of extended usage of a non-invasive passive hip exoskeleton on the quality of life of older adults. This will be achieved by analyzing the spatiotemporal gait characteristics in a feasibility study conducted over a 12-week period of consistent device usage. Additionally, the study aims to ascertain the persistence of these effects for a duration of 6 weeks post-usage.

ELIGIBILITY:
Inclusion Criteria:

* score of ≤ 5 on the Tilburg Frailty index
* able to walk independently without walking aids.

Exclusion Criteria:

* score of >6 on the Tilburg Frailty index
* uncorrected visual or hearing impairments
* Vestibular dysfunctions
* current use of walking aids.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Walking speed | Pre-test (baseline) initial, 4-weeks evaluation, 12-weeks (end of intervention) and 6-weeks post-test subsequent the 12- week intervention trial
  Changes in speed (m/s) will be assessed 1) with and without the exoskeleton 2) will be assessed through 1) a 6-minutes' walk test and 2) a short performance battery test using an inertial measurement unit (IMU) located on the fifth lumbar vertebra (L5).
Step length | Pre-test (baseline) initial, 4-weeks evaluation, 12-weeks (end of intervention) and 6-weeks post-test subsequent the 12- week intervention trial
  Changes in step length (cm) will be assessed 1) with and without the exoskeleton 2) will be assessed through 1) a 6-minutes' walk test and 2) a short performance battery test using an inertial measurement unit (IMU) located on the fifth lumbar vertebra (L5).
Double support time | Pre-test (baseline) initial, 4-weeks evaluation, 12-weeks (end of intervention) and 6-weeks post-test subsequent the 12- week intervention trial
  Changes in double support time (s) will be assessed 1) with and without the exoskeleton 2) will be assessed through 1) a 6-minutes' walk test and 2) a short performance battery test using an inertial measurement unit (IMU) located on the fifth lumbar vertebra (L5).
Cadence | Pre-test (baseline) initial, 4-weeks evaluation, 12-weeks (end of intervention) and 6-weeks post-test subsequent the 12- week intervention trial
  Changes in cadence (steps/minute) will be assessed 1) with and without the exoskeleton 2) will be assessed through 1) a 6-minutes' walk test and 2) a short performance battery test using an inertial measurement unit (IMU) located on the fifth lumbar vertebra (L5).

SECONDARY OUTCOMES:
Heart rate | Pre-test (baseline) initial, 4-weeks evaluation, 12-weeks (end of intervention) and 6-weeks post-test subsequent the 12- week intervention trial
  using a chest strap device which will be monitored during the gait measurement
Perceived effort | Pre-test (baseline) initial, 4-weeks evaluation, 12-weeks (end of intervention) and 6-weeks post-test subsequent the 12- week intervention trial
  assessed using Borg Category-Ratio (CR) scale (0 = No effort, 10 = Maximal effort) to evaluate the work tasks conducted during the pre- and post-tests.
Physical activity levels | Pre-test (baseline) initial, 4-weeks evaluation, 12-weeks (end of intervention) and 6-weeks post-test subsequent the 12- week intervention trial
  assessed using a questionnaire (The International Physical Activity Questionnaire) to determine the kind and level of the physical activity performed within the past 7 days. The questionnaire will be applied at baseline and every week for the entire duration of the intervention.
Self-reporting of exoskeleton-use during the 12-weeks intervention | Pre-test (baseline) initial, 4-weeks evaluation, 12-weeks (end of intervention) and 6-weeks post-test subsequent the 12- week intervention trial
  assessed using yes/ no, metric and open-ended questions on usage: Q1: "Did you wear the device this week?", Q2: "How much did you wear the device every day? " Q3: "What activities did you predominately performed with the device?". The questionnaire will be applied at baseline and every week for the entire duration of the intervention.
Wearability | Pre-test (baseline) initial, 4-weeks evaluation, 12-weeks (end of intervention) and 6-weeks post-test subsequent the 12- week intervention trial
  assessed using yes/ no and open-ended questions on ease/discomfort of wearing the device: Q1: "Did you have any technical problems with the device broken/stuck?" Q2: "Did you have any physical problems with the device pain/discomfort?" Q3: "Did see or feel any improvements in your ability to walk?" 4. "How would you describe your experience so far in few words? ". The questionnaire will be applied at baseline and every week for the entire duration of the intervention.
Qualitative data | Pre-test (baseline) initial, 4-weeks evaluation, 12-weeks (end of intervention) and 6-weeks post-test subsequent the 12- week intervention trial.]
  Assessed using a semi-constructed interview with yes/ no and open-ended questions on the overall experience of using the device.
Acceptability | Pre-test (baseline) initial, 4-weeks evaluation, 12-weeks (end of intervention) and 6-weeks post-test subsequent the 12- week intervention trial
  of incorporating a passive assistive bilateral exoskeleton into the daily routine of pre-frail adults for a duration of 12-weeks using the acceptability questionnaire that has a 7-point Liker scale ranging from "very unacceptable" to "very acceptable".
Life quality | Pre-test (baseline) initial, 4-weeks evaluation, 12-weeks (end of intervention) and 6-weeks post-test subsequent the 12- week intervention trial
  assessed using a questionnaire the EQ-5D-5L which evaluates five dimensions (mobility, self-care, usual activities, pain and discomfort, anxiety, and discomfort) at five severity levels ranging from no effect/symptom to slightly, moderate, severe, and extreme.
Age | Pre-test (baseline) initial, 4-weeks evaluation, 12-weeks (end of intervention) and 6-weeks post-test subsequent the 12- week intervention trial
  will be collected as descriptive statistics and for the inclusion criteria.
BMI | Pre-test (baseline) initial, 4-weeks evaluation, 12-weeks (end of intervention) and 6-weeks post-test subsequent the 12- week intervention trial
  will be assessed by collecting weigth and height.
Frailty | Pre-test (baseline) initial, 4-weeks evaluation, 12-weeks (end of intervention) and 6-weeks post-test subsequent the 12- week intervention trial
  assessed using a questionnaire the Tilburg Frailty Index which evaluates frailty levels for the inclusion criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina-Ioana Pirscoveanu, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Gistrup, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andreasen J, Lund H, Aadahl M, Gobbens RJ, Sorensen EE. Content validation of the Tilburg Frailty Indicator from the perspective of frail elderly. A qualitative explorative study. Arch Gerontol Geriatr. 2015 Nov-Dec;61(3):392-9. doi: 10.1016/j.archger.2015.08.017. Epub 2015 Aug 24. PMID 26323651
- [Background] Asselin P, Knezevic S, Kornfeld S, Cirnigliaro C, Agranova-Breyter I, Bauman WA, Spungen AM. Heart rate and oxygen demand of powered exoskeleton-assisted walking in persons with paraplegia. J Rehabil Res Dev. 2015;52(2):147-58. doi: 10.1682/JRRD.2014.02.0060. PMID 26230182
- [Background] Bangsbo J, Blackwell J, Boraxbekk CJ, Caserotti P, Dela F, Evans AB, Jespersen AP, Gliemann L, Kramer AF, Lundbye-Jensen J, Mortensen EL, Lassen AJ, Gow AJ, Harridge SDR, Hellsten Y, Kjaer M, Kujala UM, Rhodes RE, Pike ECJ, Skinner T, Skovgaard T, Troelsen J, Tulle E, Tully MA, van Uffelen JGZ, Vina J. Copenhagen Consensus statement 2019: physical activity and ageing. Br J Sports Med. 2019 Jul;53(14):856-858. doi: 10.1136/bjsports-2018-100451. Epub 2019 Feb 21. PMID 30792257
- [Background] Brustio PR, Magistro D, Zecca M, Rabaglietti E, Liubicich ME. Age-related decrements in dual-task performance: Comparison of different mobility and cognitive tasks. A cross sectional study. PLoS One. 2017 Jul 21;12(7):e0181698. doi: 10.1371/journal.pone.0181698. eCollection 2017. PMID 28732080
- [Background] Chen B, Zi B, Qin L, Pan Q. State-of-the-art research in robotic hip exoskeletons: A general review. J Orthop Translat. 2019 Oct 14;20:4-13. doi: 10.1016/j.jot.2019.09.006. eCollection 2020 Jan. PMID 31908928
- [Background] Collins SH, Wiggin MB, Sawicki GS. Reducing the energy cost of human walking using an unpowered exoskeleton. Nature. 2015 Jun 11;522(7555):212-5. doi: 10.1038/nature14288. Epub 2015 Apr 1. PMID 25830889
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Khosravi P, Ghapanchi AH. Investigating the effectiveness of technologies applied to assist seniors: A systematic literature review. Int J Med Inform. 2016 Jan;85(1):17-26. doi: 10.1016/j.ijmedinf.2015.05.014. Epub 2015 Jun 11. PMID 26216463
- [Background] Lange-Maia BS, Newman AB, Strotmeyer ES, Harris TB, Caserotti P, Glynn NW. Performance on fast- and usual-paced 400-m walk tests in older adults: are they comparable? Aging Clin Exp Res. 2015 Jun;27(3):309-14. doi: 10.1007/s40520-014-0287-y. Epub 2014 Nov 6. PMID 25373610
- [Background] Lee SH, Lee HJ, Chang WH, Choi BO, Lee J, Kim J, Ryu GH, Kim YH. Gait performance and foot pressure distribution during wearable robot-assisted gait in elderly adults. J Neuroeng Rehabil. 2017 Nov 28;14(1):123. doi: 10.1186/s12984-017-0333-z. PMID 29183379
- [Background] McPhee JS, French DP, Jackson D, Nazroo J, Pendleton N, Degens H. Physical activity in older age: perspectives for healthy ageing and frailty. Biogerontology. 2016 Jun;17(3):567-80. doi: 10.1007/s10522-016-9641-0. Epub 2016 Mar 2. PMID 26936444
- [Background] Mundt M, Batista JP, Markert B, Bollheimer C, Laurentius T. Walking with rollator: a systematic review of gait parameters in older persons. Eur Rev Aging Phys Act. 2019 Sep 10;16:15. doi: 10.1186/s11556-019-0222-5. eCollection 2019. PMID 31528238
- [Background] Panizzolo FA, Bolgiani C, Di Liddo L, Annese E, Marcolin G. Reducing the energy cost of walking in older adults using a passive hip flexion device. J Neuroeng Rehabil. 2019 Oct 15;16(1):117. doi: 10.1186/s12984-019-0599-4. PMID 31615535
- [Background] Sawicki GS, Beck ON, Kang I, Young AJ. The exoskeleton expansion: improving walking and running economy. J Neuroeng Rehabil. 2020 Feb 19;17(1):25. doi: 10.1186/s12984-020-00663-9. PMID 32075669
- [Background] Shin CN, Lee YS, Belyea M. Physical activity, benefits, and barriers across the aging continuum. Appl Nurs Res. 2018 Dec;44:107-112. doi: 10.1016/j.apnr.2018.10.003. Epub 2018 Oct 17. PMID 30389054
- [Background] Tramontano M, Morone G, Curcio A, Temperoni G, Medici A, Morelli D, Caltagirone C, Paolucci S, Iosa M. Maintaining gait stability during dual walking task: effects of age and neurological disorders. Eur J Phys Rehabil Med. 2017 Feb;53(1):7-13. doi: 10.23736/S1973-9087.16.04203-9. Epub 2016 Aug 30. PMID 27575014
- [Background] Villumsen M, Grarup B, Christensen SWMP, Palsson TS, Hirata RP. "Study protocol for the >/=65 years NOrthern jutland Cohort of Fall risk Assessment with Objective measurements (the NOCfao study)". BMC Geriatr. 2020 Jun 8;20(1):198. doi: 10.1186/s12877-020-01535-6. PMID 32513121
- [Background] Witte KA, Fiers P, Sheets-Singer AL, Collins SH. Improving the energy economy of human running with powered and unpowered ankle exoskeleton assistance. Sci Robot. 2020 Mar 25;5(40):eaay9108. doi: 10.1126/scirobotics.aay9108. PMID 33022600
- [Background] Yandell MB, Tacca JR, Zelik KE. Design of a Low Profile, Unpowered Ankle Exoskeleton That Fits Under Clothes: Overcoming Practical Barriers to Widespread Societal Adoption. IEEE Trans Neural Syst Rehabil Eng. 2019 Apr;27(4):712-723. doi: 10.1109/TNSRE.2019.2904924. Epub 2019 Mar 14. PMID 30872237
- See also: Danish Health Authority. Health promotion package - Physical activity. (2018). — https://www.sst.dk/-/media/English/Publications/2020/Forebyggelsepakke-fysisk-aktivitet-(Engelsk)/Health-promotion-package-on-physical-activity.ashx?sc_lang=en&hash=F3BB1EEB328D772F7DD3A4DF4E9B6866
- See also: Sundhedsstyrelsen. Danskernes Sundhed - Tal fra Den Nationale Sundhedsprofil — https://www.danskernessundhed.dk
- See also: World Health Organization. Denmark Physical activity factsheet 2018 — https://www.euro.who.int/__data/assets/pdf_file/0008/382373/denmark-eng.pdf
- See also: Zhang et al., 2019 - Design and Control of a Series Elastic Actuator With Clutch for Hip Exoskeleton for Precise Assistive Magnitude and Timing Control and Improved Mechanical Safety — https://ieeexplore.ieee.org/stamp/stamp.jsp?arnumber=8782586